CLINICAL TRIAL: NCT04779385
Title: Cost and Effectiveness of Pressurized Intraperitoneal Aerosol Chemotherapy (PIPAC) in Patients With Peritoneal Carcinoma.
Brief Title: Cost and Effectiveness of Pressurized Intraperitoneal Aerosol Chemotherapy in Patients With Peritoneal Carcinoma.
Acronym: PIPAC-GRE
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: CHUGA
Record Dates: First submitted 2021-02-26; First posted 2021-03-03 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-02

CONDITIONS: Evaluate the Cost of a PIPAC Procedure and the Associated Hospital Stay in France

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: PIPAC — under general anaesthesia, a laparoscopy was performed using an open laparoscopic technique to prevent intestinal wounds, which would contraindicate the procedure. A 12 mmHg pneumoperitoneum was created, and to ensure the safety of the procedure the pressure of the pneumoperitoneum was maintained constant throughout the procedure. Two laparoscopic balloon trocars (of 11 and 12 mm) were used. A thorough exploration of the abdomen, Peritoneal Cancer Index assessment, images, peritoneal biopsies, and ascites cytology (in the case of ascites) were performed prior to administration of the chemotherapy aerosol.
  For carcinomas of gastric origin, Doxurubicin at a dose of 1.5 mg/m2 was administered in combination with Cisplatin 7.5 mg/m2 diluted in 40 and 150 mL of 0.9% sodium chloride, respectively. In the case of contraindication, Oxaliplatine at a dose of 92 mg/m2 in a 5% dextrose solution was recommended.

SUMMARY:
The presence of peritoneal carcinomatosis indicates a neoplastic disease evolved. Without intervention, the prognosis is poor with survival of only a few months. Standard treatment is based on systemic chemotherapy, however, the pharmacokinetics of drug delivery to the peritoneum is poor, with limited efficacy compared to other metastatic sites such as the liver or lung. When the carcinomas are is resectable, selected patients can benefit from targeted therapeutic approaches combining peritonectomy and Hyperthermic Intraperitoneal Chemotherapy (HIPEC), offering a significant improvement in survival. A new surgical technique has been developed for patients with unresectable Chemotherapy intraperitoneal aerosol spray (PIPAC). The objective is to improve the survival time, quality of life but can also make PC resectable and therefore accessible to complete excisional surgery. The cost of this treatment is not yet fully assessed in France. The main objective of this study is to assess the real cost of PIPAC in order to allow its dissemination.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Patients treated with PIPAC and monitored for peritoneal carcinoma
* Patients informed

Exclusion Criteria:

* Patients opposition

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with peritoneal carcinomatosis of any origin treated with PIPAC.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Evaluate the cost of a PIPAC | 90 Days
  Evaluate the cost of a PIPAC procedure and the associated hospital stay

CONTACTS AND LOCATIONS:
Locations (1):
- CHUGA, Grenoble, France

IPD SHARING:
Plan to Share IPD: No